CLINICAL TRIAL: NCT02563860
Title: Pharmacological Treatment of Rett Syndrome With 3-Hydroxy-3 Methylglutaryl-coenzyme A Reductase Inhibitor-Lovastatin (Mevacor)
Brief Title: Pharmacological Treatment of Rett Syndrome With Statins
Acronym: Statins
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Rett Syndrome Research Trust (Other)
Responsible Party: Principal Investigator, Aleksandra Djukic, Professor of Clinical Neurology, Director, Tri State Rett Syndrome Center, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-4253
Record Dates: First submitted 2015-07-20; First posted 2015-09-30 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Rett Syndrome
Keywords: Treatment trial; Lovastatin
MeSH Terms: conditions — Rett Syndrome | interventions — Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental): Treatment with Lovastatin, dose escalating trial according to the following schedule:
  10 mg daily for 8 week 20 mg daily for 8 weeks 40 mg daily for 16 weeks.
  Interventions: Drug: Lovastatin

INTERVENTIONS:
Drug: Lovastatin — dose escallating
  Other Names: Mevacor

SUMMARY:
This is a phase 2 , open label, dose escalating study of Lovastatin in Rett syndrome.

DETAILED DESCRIPTION:
Excess neuronal cholesterol plays a role in the pathophysiology of Rett syndrome(RTT) and the investigators hypothesise that inhibition of cholesterol synthesis in the CNS will reduce neuronal cholesterol and lead to improvement in Rett syndrome related symptoms.

Goal: To determine the optimal dosing regiment of Lovastatin for patients with RTT and to identify the most appropriate primary outcome measure for the subsequent Phase 3 study.

Phase 2, dose escalation study.

Primary outcome: Gait speed Secondary outcomes: respiratory function, cognition, EEG (encephalopathy), Rett syndrome severity scale, neurodevelopmental assessment (QOL)

20 ambulatory female patients with genetically confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Females patients,
* Genetically confirmed RTT,
* Ambulatory.

Exclusion Criteria:

* Presence of co morbid non-Rett related disease,
* History of adverse reaction/hypersensitivity to statins,
* Levels of aspartate-amino trans-ferase (AST), alanine-amino transferase (ALT) or creatine kinase (CK) triple the normal values,
* Active liver disease,
* Concomitant use of strong CYP3A4 inhibitors,
* Condition predis-posing to renal failure secondary to rhabdomyolysis (scoliosis surgery within 6 months),
* Oral contraceptives use.

Min Age: 3 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Djukic, MD PhD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label: Treatment with Lovastatin, dose escalating trial according to the following schedule:
  All participants were assigned to the specified sequence of interventions and all participants received all the three dosing regimen please make this explicit in the Arm/Group Description. In either case, separate Period 1-10 mg daily for 8 week Period 2-20 mg daily for 8 weeks Period 3-40 mg daily for 16 weeks.
  Lovastatin: dose escallating
Period: Overall Study
Arm/Group | Open Label
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Open Label: Female patients with genetically confirmed RTT, treatment arm only.
  Treatment with Lovastatin, dose escalating trial according to the following schedule:
  10 mg daily for 8 week 20 mg daily for 8 weeks 40 mg daily for 16 weeks.
  Lovastatin: dose escallating
Arm/Group | Open Label
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Gait Velocity as Measured by GAITRite System
Description: To perform quantitative gait assessment using a computerized walkway with embedded pressure sendors (GAIT rite)
Time Frame: During final week of treatment, week 32
Measure: Median (Inter-Quartile Range); unit: cm/sec
Groups:
- Open Label: Treatment with Lovastatin, dose escalating trial according to the following schedule:
  10 mg daily for 8 week 20 mg daily for 8 weeks 40 mg daily for 16 weeks.
  Lovastatin: dose escallating
Arm/Group | Open Label
Number analyzed (Participants) | 19
cm/sec | 58.6 [43.8 to 71.1]

2. Secondary Outcome: Visual Memory Novelty Score as Assessed by TobiiTX 300 Eyetracking System
Description: Novelty score is considered a composite measure of visual memory.Test is a standardized neuropsychological test( "Rose test") adapted for eye tracking system.
  The present study made use of a well-established battery of "visual paired comparison" problems .There were nine problems: five using achromatic photos of faces and four using multicolored abstract patterns paired stimuli , separated by 23°. For each problem, two identical stimuli are briefly presented side by side for familiarization, then the familiar and a new one are paired on test
  Recognition(memory) is indexed by a novelty score (percentage of looking to the novel target on test).
  Higher novelty scores were related to better recognition (index of better memory) Scores range from 0.0-1.0 (0-100%) and indicate 1) more overall looking at novel target and (2) more fixations to novel targets.
  Score of .5 (50%) indicates looking "by change" only with no recognition.
Time Frame: final week of treatment, Week 32
Population: Calculation done on intent-to-treat population
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Open Label
Number analyzed (Participants) | 19
percent
  Pre-treatment | 44.85 [25.85 to 68.10]
  Post treatment | 58.93 [47.55 to 70.25]

ADVERSE EVENTS:
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=20)
mild (Psychiatric disorders) | 1 (1) — Anxiety, upon dose escalation from 20 to 40 mg of Lovastatin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No